CLINICAL TRIAL: NCT01297491
Title: An Open Label Two-stage Study of Orally Administered BKM120 in Patients With Metastatic Non-small Cell Lung Cancer With Activated PI3K Pathway
Brief Title: Safety and Efficacy of BKM120 in Patients With Metastatic Non-small Cell Lung Cancer
Acronym: BASALT-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CBKM120D2201; 2010-024011-14 (EudraCT Number)
Record Dates: First submitted 2011-02-11; First posted 2011-02-16 (Estimated); Results first posted 2016-02-02 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; PI3K
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Squamous BKM120 100mg qd (Experimental): Diagnosed patients with non-small cell lung cancer (NSCLC) that progressed after one prior, platinum-based chemotherapy line for metastatic disease.
  Interventions: Drug: BKM120
- Non-Squamous BKM120 100mg qd (Experimental): Diagnosed patients with non-squamous NSCLC that progressed after one or two prior antineoplastic therapy lines for metastatic disease.
  Interventions: Drug: BKM120

INTERVENTIONS:
Drug: BKM120 — Buparlisib was supplied as 10mg or 50mg capsules. It was administered on a continuous once daily dosing schedule at a dose of 100 mg. The patient was dosed on a flat scale of mg/day and not adjusted to body weight or body surface area.
  Other Names: Buparlisib

SUMMARY:
The purpose of this two-stage phase II study is to assess the efficacy of BKM120, as measured by determining the progression free survival (PFS), in patients with pretreated metastatic Non-small Cell Lung Cancer (NSCLC) that exhibits PI3K pathway activation. BKM120 will be investigated in two groups of NSCLC patients according to the histology of the cancer: squamous and non-squamous.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC with activated PI3K pathway
* Progressive disease after prior systemic antineoplastic treatment(s) for advanced NSCLC
* Archival or fresh tumor biopsy must be available for profiling
* Measurable and/or non-measurable disease as per RECIST 1.1 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Adequate organ function as assessed by laboratory tests

Exclusion Criteria:

* Patient has received previous treatment with PI3K inhibitors
* Patient with squamous NSCLC has received more than one line of chemotherapy treatment for metastatic disease; patient with non-squamous NSCLC has received more than two lines of systemic antineoplastic treatment for metastatic disease
* Uncontrolled or symptomatic CNS metastases
* Concurrent use of any other approved or investigational antineoplastic agent
* Radiotherapy ≤ 28 days prior to starting study drug
* Major surgery within 28 days prior to starting study drug
* History of clinically significant cardiac dysfunction, mood disorders, or poorly controlled diabetes mellitus
* Current treatment with medication that has a known risk to prolong the QT interval or inducing Torsades de Pointes
* Impairment of gastrointestinal (GI) function
* Chronic treatment with steroids or another immunosuppressive agent.
* Concurrent severe and/or uncontrolled medical condition
* Currently receiving Warfarin or another coumarin derivative
* Known history of HIV infection
* Sensory neuropathy with functional impairment (CTC grade 2 neuropathy, regardless of causality)
* Pregnancy, lactation, or breastfeeding
* Woman of child-bearing potential

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2011-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (90):
- United States (32):
  - Ironwood Cancer and Research Centers SC, Chandler, Arizona
  - Arizona Oncology Associates Tucson (Rudasill & La Cholla), Phoenix, Arizona
  - Mayo Clinic - Arizona Mayo Scottsdale AZ, Scottsdale, Arizona
  - Highlands Oncology Group Dept of Highlands Oncology Grp, Fayetteville, Arkansas
  - Cedars Sinai Medical Center Dept.of Cedars-Sinai Med. Ctr., Los Angeles, California
  - University of California at San Diego, Moores Cancer Ctr SC, San Diego, California
  - University of Colorado Univ CO, Aurora, Colorado
  - Rocky Mountain Cancer Centers Dept. of Rocky Mountain Cancer, Greenwood Village, Colorado
  - H. Lee Moffitt Cancer Center & Research Institute H Lee Moffitt, Tampa, Florida
  - Emory University School of Medicine/Winship Cancer Institute Emory 2, Atlanta, Georgia
  - Rush University Medical Center SC, Chicago, Illinois
  - University of Chicago Medical Center Unvi Chi, Chicago, Illinois
  - University of Kansas Cancer Center Univ of KS, Kansas City, Kansas
  - Massachusetts General Hospital Mass General, Boston, Massachusetts
  - Fallon Clinic at Worcester Medical Center Fallon Clinic Worcester Med, Worcester, Massachusetts
  - Karmanos Cancer Institute Wayne St Karmanos, Detroit, Michigan
  - Washington University School of Medicine Washington University (16), St Louis, Missouri
  - Hematology Oncology Associates of Northern New Jersey PA DeptofHem-OncofNorthern NJ (2), Morristown, New Jersey
  - Overlook Hospital - Carol G Simon Cancer Center Carol G Simon, Summit, New Jersey
  - Roswell Park Cancer Institute Rosewell, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center Sloan Kettering, New York, New York
  - Duke University Medical Center Duke 2, Durham, North Carolina
  - MetroHealth Medical Center Dept.ofMetroHealthMedCtr.(2), Cleveland, Ohio
  - University of Oklahoma Health Sciences Center Dept. of Oklahoma Univ. HSC, Oklahoma City, Oklahoma
  - Northwest Cancer Specialists Compass Oncology -BKM, Portland, Oregon
  - University of Pittsburgh Medical Center SC-2, Pittsburgh, Pennsylvania
  - Medical University of South Carolina MUSC, Charleston, South Carolina
  - Baylor Health Care System/Sammons Cancer Center Baylor Texas Oncology, Dallas, Texas
  - Texas Oncology South Texas Oncology, Dallas, Texas
  - U of TX Southwestern Medical Center - SimmonsCompCancerCtr Clinical Research Office, Dallas, Texas
  - Virginia Oncology Associates VOA - Lake Wright (2), *see Various Departments*, Virginia
  - University of Wisconsin Univ WIsc 2, Madison, Wisconsin
- Argentina (3):
  - Novartis Investigative Site, Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Córdoba, Córdoba Province
  - Novartis Investigative Site, Rio Negro, Viedma
- Belgium (5):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Charleroi
  - Novartis Investigative Site, Genk
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Libramont
- Brazil (5):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Florianópolis, Santa Catarina
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (3):
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- France (5):
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Villejuif
- Germany (9):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Nuremberg
  - Novartis Investigative Site, Oldenburg
  - Novartis Investigative Site, Recklinghausen
- Novartis Investigative Site, Hong Kong, Hong Kong
- Hungary (4):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Deszk
  - Novartis Investigative Site, Mátraháza
  - Novartis Investigative Site, Szolnok
- Italy (5):
  - Novartis Investigative Site, Avellino, AV
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Udine, UD
- Japan (2):
  - Novartis Investigative Site, Kurashiki, Okayama-ken
  - Novartis Investigative Site, Koto, Tokyo
- Novartis Investigative Site, Maastricht, Netherlands
- Novartis Investigative Site, Singapore, Singapore, Singapore
- Spain (4):
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Mataró, Catalonia
  - Novartis Investigative Site, Alicante, Valencia
- Taiwan (2):
  - Novartis Investigative Site, Tainan, Taiwan ROC
  - Novartis Investigative Site, Taipei, Taiwan ROC
- Thailand (2):
  - Novartis Investigative Site, Bangkok
  - Novartis Investigative Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Izmir, Turkey
  - Novartis Investigative Site, Altunizade
- United Kingdom (4):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Leicester
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester

REFERENCES:
- [Result] Vansteenkiste JF, Canon JL, De Braud F, Grossi F, De Pas T, Gray JE, Su WC, Felip E, Yoshioka H, Gridelli C, Dy GK, Thongprasert S, Reck M, Aimone P, Vidam GA, Roussou P, Wang YA, Di Tomaso E, Soria JC. Safety and Efficacy of Buparlisib (BKM120) in Patients with PI3K Pathway-Activated Non-Small Cell Lung Cancer: Results from the Phase II BASALT-1 Study. J Thorac Oncol. 2015 Sep;10(9):1319-1327. doi: 10.1097/JTO.0000000000000607. PMID 26098748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Started | 30 | 33
Completed | 0 | 0
Not Completed | 30 | 33
Not completed — Adverse Event | 11 | 6
Not completed — Physician Decision | 3 | 2
Not completed — Progressive disease | 11 | 20
Not completed — Patient/Guardian decision | 3 | 4
Not completed — Death | 2 | 1

BASELINE CHARACTERISTICS:
Population: Analysis set Stage 1 includes all patients who were enrolled during Stage 1 after meeting eligibility criteria and who have received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Customized [Number; unit: Participants]
  < 65 years | 12 | 19 | 31
  >= 65 years | 18 | 14 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 14 | 23
  Male | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) Rate as Per Investigator Local Review Measured Using RECIST 1.1 of Patients at Week 12
Description: PFS rate was defined as the percentage of participants who were progression free at 12 weeks. Participants were considered as a "success" for PFS rate evaluated at 12 weeks if they presented an overall response at their 2nd post-baseline tumor assessment.The enrollment into the study in either histology group would stop for futility if a PFS rate <50% at 12 weeks was observed.
  No statistical analysis was planned for this primary outcome. The results of the primary objective was based on the data from the interim analysis that took place at the cut off dates: 10-Apr-2013 for non-squamous and 08-Jan-2014 for squamous group.
Time Frame: Week 12
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Number analyzed (Participants) | 30 | 30
Percentage of participants | 23.3 [9.9 to 42.3] | 20.0 [7.7 to 38.6]

2. Secondary Outcome: Overall Survival (OS) Using Kaplan-Meier Estimates
Description: OS was defined as the time from start of study drug (Stage 1) until death from any cause. If a patient was not known to have died, survival was censored at the date of last contact.
Time Frame: Every 8 weeks up to 24 months
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Number analyzed (Participants) | 30 | 33
Months | 7.98 [5.95 to 10.09] | 7.20 [4.01 to 9.92]

3. Secondary Outcome: Overall Response Rate (ORR) Based on Investigator Assessment
Description: ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR). Complete response was defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. Partial response was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Analyses of response rates were performed based on investigators' assessments (as per RECIST 1.1 criteria). ORR included all patients with and without measurable disease at baseline.
Time Frame: Every 6 weeks up to 24 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Number analyzed (Participants) | 30 | 33
Percentage of participants | 3.3 | 3.0

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR defined as the percentage of participants with best overall response of CR or PR or stable disease (SD). Complete response was defined as disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm. Partial response was defined as at least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters. Stable Disease (SD): Neither sufficient shrinkage to qualify for PR or CR nor an increase in lesions which would qualify for PD.
  Analyses of response rates were performed based on investigators' assessments (as per RECIST 1.1 criteria). DCR included all participants with and without measurable disease at baseline.
Time Frame: Every 6 weeks up tp 24 months
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Number analyzed (Participants) | 30 | 33
Percentage of participants | 46.7 | 45.5

5. Secondary Outcome: Time to Response (TTR)
Description: TTR for a participant was defined as the time from the first treatment date to the date of first documented confirmed CR or PR evaluation. The date of event was defined as the date of response that was first determined and not using the date the response was confirmed.
Time Frame: Every 6 weeks up to 24 months
Population: Analysis set Stage 1 includes all patients who were enrolled during Stage 1 after meeting eligibility criteria and who have received at least 1 dose of study drug. 1 partial response was observed as best overall response (BOR) for 1 patient in the squamous group. Also,1 patient experienced partial response as BOR in the non-squamous group.
Measure: Number; unit: Days
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Number analyzed (Participants) | 30 | 33
Days | 41 | 42

6. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined as the elapsed time between the date of first documented CR or PR response (not the date of confirmed response) and the following date of event defined as the first documented progression or death due to underlying cancer.
Time Frame: Every 6 weeks up to 24 months
Population: as for outcome 5
Measure: Number; unit: Days
Arm/Group | Squamous BKM120 100mg qd | Non-Squamous BKM120 100mg qd
Number analyzed (Participants) | 30 | 33
Days | 73 | 85

ADVERSE EVENTS:
Groups:
- Squamous BKM120 100 mg qd: Diagnosed patients with non-small cell lung cancer (NSCLC) that progressed after one prior, platinum-based chemotherapy line for metastatic disease.
- Non-Squamous BKM120 100 mg qd: Diagnosed patients with non-squamous NSCLC that progressed after one or two prior antineoplastic therapy lines for metastatic disease.
Arm/Group | Squamous BKM120 100 mg qd | Non-Squamous BKM120 100 mg qd
Serious Adverse Events (participants affected / at risk) | 16/30 | 15/33
Other Adverse Events (participants affected / at risk) | 29/30 | 32/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Squamous BKM120 100 mg qd (N=30) | Non-Squamous BKM120 100 mg qd (N=33)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiogenic shock (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Blepharitis (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 4 | 0
Local swelling (General disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Squamous BKM120 100 mg qd (N=30) | Non-Squamous BKM120 100 mg qd (N=33)
Anaemia (Blood and lymphatic system disorders) | 5 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0
Sinus tachycardia (Cardiac disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 2
Lacrimation increased (Eye disorders) | 2 | 1
Vision blurred (Eye disorders) | 3 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 5 | 3
Diarrhoea (Gastrointestinal disorders) | 11 | 11
Dry mouth (Gastrointestinal disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 13 | 9
Stomatitis (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 6 | 5
Asthenia (General disorders) | 6 | 12
Fatigue (General disorders) | 11 | 6
Hypothermia (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 3 | 1
Oedema peripheral (General disorders) | 3 | 1
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 4
Bronchitis (Infections and infestations) | 4 | 0
Candida infection (Infections and infestations) | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 3
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Rhinitis (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 6 | 6
Aspartate aminotransferase increased (Investigations) | 5 | 6
Blood alkaline phosphatase increased (Investigations) | 3 | 1
Blood creatinine increased (Investigations) | 2 | 1
Blood glucose increased (Investigations) | 2 | 1
Blood lactate dehydrogenase increased (Investigations) | 2 | 2
Blood urea increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 3 | 2
Insulin c-peptide increased (Investigations) | 0 | 2
Transaminases increased (Investigations) | 2 | 2
Weight decreased (Investigations) | 8 | 3
Decreased appetite (Metabolism and nutrition disorders) | 11 | 12
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Dizziness (Nervous system disorders) | 2 | 1
Dysgeusia (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 4 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Myoclonus (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 2
Somnolence (Nervous system disorders) | 1 | 2
Tremor (Nervous system disorders) | 4 | 1
Anxiety (Psychiatric disorders) | 3 | 8
Confusional state (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 4 | 11
Insomnia (Psychiatric disorders) | 1 | 2
Mood altered (Psychiatric disorders) | 2 | 4
Renal failure acute (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 5
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 11 | 4
Rash (Skin and subcutaneous tissue disorders) | 8 | 6
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 2
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.